CLINICAL TRIAL: NCT06854731
Title: ACTIVE: Adding Life to Years in Cognitive Frailty by Preventing Falls
Brief Title: Preventing Falls in Older Adults With Cognitive Frailty
Acronym: ACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H23-01584
Record Dates: First submitted 2025-02-17; First posted 2025-03-03 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Falls; Frailty; Mild Cognitive Impairment
Keywords: execise; falls; cognitive frailty
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Control (Active Comparator): All active control participants will be invited to join monthly interactive education sessions via Zoom or in-person.
  Interventions: Other: Education Session
- Otago Exercise Program (OEP) Plus (Experimental): The OEP+ intervention integrates the OEP with health coaching by a physical therapists or kinesiologist. The OEP is an individualized home-based balance and strength exercise training program delivered by a PT or kinesiologist coach over 5 home visits
  Interventions: Behavioral: Balance and Strength Training Exercises with Health Coaching

INTERVENTIONS:
Behavioral: Balance and Strength Training Exercises with Health Coaching — The OEP+ intervention integrates the OEP with health coaching by a physical therapists or kinesiologist. The OEP is an individualized home-based balance and strength exercise training program delivered by a PT or kinesiologist coach over 5 home visits.
  Other Names: Otago Exercise Program Plus (OEP+)
  Arms: Otago Exercise Program (OEP) Plus
Other: Education Session — All active comparator participants will be invited to join monthly interactive social and education sessions via Zoom or in-person (hybrid delivery).
  Arms: Educational Control

SUMMARY:
The Problem: The proposed trial will address the problem of how to effectively prevent subsequent falls in community-dwelling cognitively frail older adults with a history of falls.

Primary Question: In community-dwelling older adults with cognitive frailty and a history of falls, can a home-based exercise program with behavioural change techniques significantly reduce falls vs. health education (i.e., control; CON)?

DETAILED DESCRIPTION:
Rationale: Falls are a significant cause of functional decline and often a sentinel event. Older adults with cognitive frailty - those with concurrent physical frailty and mild cognitive impairment - are at particular risk for falls. Notably, falls can cause a sudden and severe change in their health state from one of independence to one of dependence. Thus, effective falls prevention strategies need to be identified for older adults with cognitive frailty.

The Otago Exercise Program (OEP) - a physical therapist (PT) delivered home-based exercise program - is an evidence-based falls prevention program for community-dwelling older adults. Our pilot data show the OEP vs. usually care significantly reduced subsequent falls in 192 community-dwelling older adults with cognitive frailty and a history of falls; the incident rate ratio was 0.64 (95% CI, 0.43-0.98; P = .042). These preliminary findings need to be confirmed in a rigorously designed RCT powered for falls in older adults with cognitive frailty; none exist to date.

We also observed lower OEP adherence among older adults with cognitive frailty vs. those without cognitive frailty. Thus, strategies to support adherence must be considered in RCTs of exercise to prevent falls in this high-risk population. Evidence-based strategies include health coaching.

Thus, we propose a 12-month multi-site randomized controlled trial (RCT) in older adults with cognitive frailty and a history of falls to assess the efficacy of the OEP combined with health coaching (i.e., OEP+) to prevent falls.

Primary Question: In community-dwelling older adults with cognitive frailty and a history of falls, can the OEP+ significantly reduce falls vs. health education (i.e., control; CON)?

Secondary Questions: 1) What are additional benefits of the OEP+ vs. CON? 2) Do the benefits of OEP+ persist 6 months post cessation? 3) Can the OEP+ reduce falls or improve quality of life at similar or lower costs vs. CON?

Methods: A 12-month assessor-blinded, multi-site RCT, with a 6-month follow-up, in older adults, with cognitive frailty - defined by a Short Physical Performance Battery score < 9/12 and a Montreal Cognitive Assessment score between 18-25/30 - and a history of falls. Participants will be randomized to either: a) OEP+ or b) CON. The OEP+ intervention will include Brief Action Planning-based health coaching. The CON group will include monthly interactive education sessions via Zoom. Measurement will occur at baseline, 6, 12, and 18 months, with falls tracked daily.

ELIGIBILITY:
Inclusion Criteria:

* We will include individuals who: 1) are aged 70 to 89 years*; 2) live in Greater Vancouver; 3) are community-dwelling (i.e., not residing in a nursing home or extended care unit); 4) experienced a non-syncopal fall in the prior 12 months; 5) scored < 9/12 on the SPPB; 6) have subjective cognitive complaints based on interview; 7) scored 18-25/30 on the MoCA; 8) are able to walk independently; use of cane is acceptable; 9) are able to safely engage in exercise as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+) and confirmed by their physician; 10) have internet at home; and 11) are able to provide written informed consent.

  * The age maximum of 89 was set due to the increased risk of significant adverse health outcomes cognitively frail older adults face. As this population has an increased risk of falls, functional disability with loss of independence, hospitalization, and death, setting an age maximum aims to increase the likelihood that participants will be able to complete the 18-month study without interruptions due to health complications. This age limit has been reviewed and approved by CIHR.

Exclusion Criteria:

* We will exclude those who are: 1) diagnosed with dementia, as measured by a Clinical Dementia Rating (CDR) score above 0.5, a neurodegenerative disease, or stroke; 2) self-report engaging in strength training and/or balance training exercises > 2 times per week, in the prior 3 months; or 3) unable to understand, speak, and read English proficiently.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Falls | Daily tracking over 12 months
  The number of self-reported falls during the 12-month intervention period (i.e., rate of falls).

SECONDARY OUTCOMES:
Short Physical Performance Battery | Baseline, 6 months, 12 months, 18 months
  A physical performance battery out of 12 points (max. performance).
Montreal Cognitive Assessment | Baseline, 6 months, 12 months, 18 months
  A test that covers multiple cognitive domains. Often used to screen for mild cognitive impairment.
Falls during followup period | Daily tracking from 12 months (trial completion) to end of 6-month followup (18 months)
  The number of self-reported falls during the 6-month ifollowup period (i.e., rate of falls).
NIH Cognitive Toolbox | Baseline, 6 months, 12 months, 18 months
  Cognitive function measured using the NIH Cognitive Toolbox
Processing speed | Baseline, 6 months, 12 months, 18 months
  Processing speed measured by Digit Symbol Substitute Test
Memory | Baseline, 6 months, 12 months, 18 months
  Memory measured by the Rey Auditory Verbal Learning Test
Gait Speed | Baseline, 6 months, 12 months, 18 months
  Walking speed in m/s measured over 4 meters (part of the Short Physical Performance Battery)
Muscle Strength | Baseline, 6 months, 12 months, 18 months
  Dominant quadriceps strength and dominant hand grip strength.
Community Mobility | Baseline, 6 months, 12 months, 18 months
  Life Space Questionnaire to measure community mobility
Functional Mobility | Baseline, 6 months, 12 months, 18 months
  Timed Up and Go Test to measure functional mobility
Fatigue | Baseline, 6 months, 12 months, 18 months
  The 9-item Fatigue Severity Scale100 will be used to assess how fatigue interferes with certain activities and its severity.
Quality of Life | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months
  The EuroQol EQ-5 Domain (5D)-5 Level (5L) (EQ-5D-5L) will assess quality of life
Fear of Falling | Baseline, 6 months, 12 months, 18 months
  Fear of falling as assessed by the Iconographical Falls Efficacy Scale (Icon-FES).
Health Resource Utilization (HRU) | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months
  Cost data will be collected every 3 months using the HRU questionnaire
Sleep Quality (Subjective) | Baseline, 6 months, 12 months, 18 months
  Sleep quality will be measured subjectively using the Pittsburgh Quality Sleep Index
Sleep Quality (Objective) - Optional | Baseline, 6 months, 12 months, 18 months
  Sleep quality parameters will be measured using ActiGraph
Brain Function - Optional | Baseline, 6 months, 12 months
  Brain function will be measured using functional near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Aging SMART at VCH, University of BC, Vancouver, British Columbia, Canada